CLINICAL TRIAL: NCT00196183
Title: Randomized Study Comparing Pulmonary Vein Isolation Alone vs. Pulmonary Vein Isolation Plus Electrogram-Guided Substrate Ablation
Brief Title: Trigger- vs. Substrate-Ablation for Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. C00504
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): trigger-guided ablation of paroxysmal atrial fibrillation
  Interventions: Procedure: trigger-guided catheter-ablation
- 2 (Experimental): trigger-+substrate guided ablation of paroxysmal atrial fibrillation
  Interventions: Procedure: trigger+substrate-guided catheter ablation

INTERVENTIONS:
Procedure: trigger-guided catheter-ablation — trigger-guided ablation of paroxysmal atrial fibrillation
  Arms: 1
Procedure: trigger+substrate-guided catheter ablation — trigger-+substrate guided ablation of paroxysmal atrial fibrillation
  Arms: 2

SUMMARY:
The purpose of this study is to compare two strategies of catheter-based treatment of paroxysmal atrial fibrillation: Pulmonary vein isolation either alone or combined with electrogram-guided substrate-ablation.

DETAILED DESCRIPTION:
Catheter ablation has evolved an accepted alternative in the curative treatment of atrial fibrillation (AF). However, discussion about the best ablation strategy is still ongoing.

In patients with paroxysmal AF, it has been reproducibly demonstrated that curing rates of approximately 65-70% can be achieved with the electric isolation of pulmonary veins (PV) eliminating the initiating triggers of AF episodes. Recently, a new catheter ablation approach targeting in both atria fractionated, complex electrograms during ongoing AF and modifying thus the substrate maintaining AF has been described. The first describer of this technique reports curing rates of 92%. We want to compare in a randomized prospective study the treatment by PV isolation alone with a combined approach of PV isolation together with ablation of fractionated complex electrograms in patients with paroxysmal AF. Study endpoint is the achievement of stable sinus rhythm as assessed by 7 days holter ECG in the absence of antiarrhythmic drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and <80 years
* Symptomatic paroxysmal atrial fibrillation
* Drug-refractory
* Anticoagulation

Exclusion Criteria:

* Hyperthyreosis
* Moderate-to-severe mitral valve valvulopathy
* LV-ejection fraction <35%
* Prior ablation, PCI or heart surgery <3 months
* Left atrial thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Sinus rhythm in follow-up in the absence of antiarrhythmic drugs after the first catheter ablation | Sinus rhythm in follow-up in the absence of antiarrhythmic drugs after the first catheter ablation

CONTACTS AND LOCATIONS:
Overall Officials: Claus Schmitt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Isabel Deisenhofer, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Background] Karch MR, Zrenner B, Deisenhofer I, Schreieck J, Ndrepepa G, Dong J, Lamprecht K, Barthel P, Luciani E, Schomig A, Schmitt C. Freedom from atrial tachyarrhythmias after catheter ablation of atrial fibrillation: a randomized comparison between 2 current ablation strategies. Circulation. 2005 Jun 7;111(22):2875-80. doi: 10.1161/CIRCULATIONAHA.104.491530. Epub 2005 May 31. PMID 15927974
- [Background] Nademanee K, McKenzie J, Kosar E, Schwab M, Sunsaneewitayakul B, Vasavakul T, Khunnawat C, Ngarmukos T. A new approach for catheter ablation of atrial fibrillation: mapping of the electrophysiologic substrate. J Am Coll Cardiol. 2004 Jun 2;43(11):2044-53. doi: 10.1016/j.jacc.2003.12.054. PMID 15172410